CLINICAL TRIAL: NCT00179387
Title: Evaluation of Mind-Body Groups on the Quality of Life of Cancer Patients
Brief Title: Mind-Body Program for Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2003-412; ACS Research Scholar's Grant
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Neoplasms
Keywords: Neoplasms; Needs Assessment; Adaptation Psychological; Minority Groups; Psychotherapy, Group; Program Evaluation; Spirituality; Spiritual Therapies
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Psycho-educational / Stress Management group
  Interventions: Behavioral: Mind-Body Psychotherapy Group
- 2 (Active Comparator): Spiritual-Existential Support Group
  Interventions: Behavioral: Mind-Body Psychotherapy Group

INTERVENTIONS:
Behavioral: Mind-Body Psychotherapy Group — Psycho-educational group
  Other Names: Stress Management Group
  Arms: 1
Behavioral: Mind-Body Psychotherapy Group — Spiritual-Existential Group
  Other Names: Spiritual Support Group
  Arms: 2

SUMMARY:
The purpose of this study is to find out if Mind-Body groups can help improve the physical and emotional well-being of people facing cancer or its treatment.

DETAILED DESCRIPTION:
Pain, fatigue, anxiety, depression, nausea, sexual impairment, body image disturbance, relationship strains, existential distress and role losses are all potential "side-effects" of living with cancer and its treatment. Behavioral interventions have shown some success in mitigating distress and QOL impairment among cancer patients. The purpose of this randomized-controlled study is to compare the effects of Mind-body group interventions on the quality of life of patients with advanced cancer. Patients are randomized to one of two psychotherapy groups, which occur weekly for eight weeks. Quality of life assessments are conducted at baseline and two and four-month intervals.

ELIGIBILITY:
Inclusion Criteria:

* On Active Treatment for:

Breast Cancer Stage IV, Colorectal Cancer Stage IV, Lung Cancer Stages III & IV, or All Other Cancers (ANY stage on treatment)

* Language is English or Spanish

Exclusion Criteria:

* Patient is currently attending other support/psychotherapy group
* Significant Cognitive Impairment
* ECOG performance status = 3 or 4
* Current major untreated psychiatric disorder
* Unable to attend intervention in following 8 weeks due to medical or practical restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2004-12-01 (Actual); Primary Completion 2016-02-25 (Actual); Study Completion 2016-02-25 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy | baseline to 2 months and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Alyson Moadel, Ph.D., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Derived] Stein EM, Kolidas E, Moadel A. Do spiritual patients want spiritual interventions?: A qualitative exploration of underserved cancer patients' perspectives on religion and spirituality. Palliat Support Care. 2015 Feb;13(1):19-25. doi: 10.1017/S1478951513000217. Epub 2013 Aug 6. PMID 23916058
- See also: Support programs for cancer patients & their families in the Bronx — http://www.einstein.yu.edu/cancercenter/support